CLINICAL TRIAL: NCT07183371
Title: A Phase IIb Randomised Controlled Trial of the Safety, Immunogenicity and Efficacy of the Malaria Vaccine Candidates R78C With Matrix-M™, and the Combination of RH5.1 and R21 With Matrix-M™, in Children Aged 5-36 Months in Burkina Faso
Brief Title: A Study to Assess the Experimental Malaria Vaccines R78C and RH5.1 With Matrix-M in Combination With R21/Matrix-M
Acronym: VAC087
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); European Vaccine Initiative (Other); Bundesministerium für Forschung, Technologie und Raumfahrt (BMFTR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAC087
Record Dates: First submitted 2025-07-02; First posted 2025-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — R21 monoclonal antibody; Matrix-M; Meningococcal Vaccines

STUDY DESIGN:
Intervention Model Description: This is a Phase IIb, double-blinded, block randomised, controlled trial to assess the safety, immunogenicity and efficacy of the blood-stage malaria vaccine candidate R78C in Matrix-M and the multi-stage combination of the blood-stage malaria vaccine candidates RH5.1 and R78C in Matrix-M and the pre-erythrocytic malaria vaccine R21 in Matrix-M.
  360 healthy children aged between 5 and 36 months at the time of first vaccination living in a malaria endemic area will be recruited at one site in Burkina Faso.
  Participants will be randomised to receive either three doses of the malaria candidate vaccines R78C/Matrix-M and three doses of a commercially available rabies vaccine, three doses of RH5.1+R78C/Matrix-M and three doses of R21/Matrix-M or six doses of commercially available control vaccines.
  Follow up will be for six months following the last vaccination.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinding will be used to reduce bias in evaluating the study endpoints. This means that the vaccine recipient, their parent(s)/guardian(s), all investigators and the study team responsible for the evaluation of efficacy, safety and immunogenicity endpoints will all be unaware of the exact treatment given to the participant. The vaccines will be different in terms of volume and colour. Therefore, the contents of the syringe will be masked with an opaque label to ensure that parent(s)/guardian(s), as well as nurse administering the vaccine are blinded.
  The central study team will remain blinded. The laboratory team involved in the immunogenicity analysis will be blinded also.
  The Local Safety Monitor (LSM) and Data Safety Monitoring Board (DSMB), will also be provided with the randomisation sequence. If deemed necessary for reasons such as safety, the LSM or DSMB will unblind the specific enrolled participant without revealing the study group to the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (n=120) children 5-36 months (Experimental): They will receive three doses of 10 µg R78C + 50 µg Matrix-M, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182). A commercially available rabies vaccine, Rabivax-S, will be administered at Month 3 (Day 98), Month 4 (Day 126) and Month 5 (Day 154). All will be given as a intramuscular injections.
  Interventions: Biological: R78C; Biological: Matrix-M™; Biological: Rabivax-S
- Group 2 (n=120) children 5-36 months (Experimental): They will receive three doses of 10 µg RH5.1 + 10 µg R78C + 50 µg Matrix-M, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182). 5 µg R21 + 50 µg Matrix-M will be administered at Month 3 (Day 98), Month 4 (Day 126) and Month 5 (Day 154), also given as Intramuscular injections. All will be given as intramuscular injections.
  Interventions: Biological: R21; Biological: RH5.1; Biological: R78C; Biological: Matrix-M™
- Group 3 (n=120) children 5-36 months (Placebo Comparator): Participants will receive six doses of commercially available control vaccines. This consists of the Hepatitis A vaccine, Avaxim 80, which will be given at Month 0 (Day 0) and Month 6 (Day 182), the meningitis vaccine, Menveo, given at Month 1 (Day 28), and a rabies vaccine, Rabivax-S, given at Month 3 (Day 98), Month 4 (Day 126) and Month 5 (Day 154). All will be given as a intramuscular injections.
  Interventions: Biological: Rabivax-S; Biological: Menveo; Biological: Avaxim 80

INTERVENTIONS:
Biological: R21 — A protein particle comprising recombinant HBsAg fused to the central repeat and the C-terminus of the circumsporozoite protein
  Arms: Group 2 (n=120) children 5-36 months
Biological: RH5.1 — A soluble protein vaccine against the RH5 antigen
  Arms: Group 2 (n=120) children 5-36 months
Biological: R78C — A soluble RIPR EGF-CyRPA fusion protein vaccine
  Arms: Group 1 (n=120) children 5-36 months; Group 2 (n=120) children 5-36 months
Biological: Matrix-M™ — A saponin-based vaccine adjuvant
  Arms: Group 1 (n=120) children 5-36 months; Group 2 (n=120) children 5-36 months
Biological: Rabivax-S — Rabivax-S is an inactivated, freeze-dried, single-dose vaccine. The vaccine contains purified, inactivated rabies antigen produced using Vero ATCC CCL 81 cells as the cell substrate, Pitman Moore (PM3218) as the virus strain, and sucrose, glycine and HSA (Human Serum Albumin) as excipients
  Arms: Group 1 (n=120) children 5-36 months; Group 3 (n=120) children 5-36 months
Biological: Menveo — Menveo is a tetravalent meningitis vaccine that consists of one vial of MenA powder and one vial of Men CWY solution.
  Arms: Group 3 (n=120) children 5-36 months
Biological: Avaxim 80 — Avaxim 80 is an inactivated, adsorbed hepatitis A vaccine. Each immunising dose contains 80 antigen units of inactivated hepatitis A virus (GBM strain).
  Arms: Group 3 (n=120) children 5-36 months

SUMMARY:
This is a Phase IIb randomised controlled trial of the safety, immunogenicity and efficacy of the malaria vaccine candidates R78C with Matrix-M™, and the combination of RH5.1 and R21 with Matrix-M™, in children aged 5-36 months in Burkina Faso.

DETAILED DESCRIPTION:
There will be three study groups, each comprising of 120 children aged between 5 and 36 months at the time of first vaccination living in a malaria endemic area and will be recruited at one site in Burkina Faso. Participants will be randomised to receive either three doses of the malaria candidate vaccines R78C/Matrix-M and three doses of a commercially available rabies vaccine, three doses of RH5.1+R78C/Matrix-M and three doses of R21/Matrix-M or six doses of commercially available control vaccines.

Follow up will be for six months following the last vaccination.

ELIGIBILITY:
Inclusion Criteria: Only participants who meet all the inclusion criteria will be enrolled into the trial:

* Healthy infant aged 5-36 months at the time of first study vaccination
* Parent/guardian provides signed/thumb-printed informed consent
* Infant and parent/guardian resident in the study area villages and anticipated to be available for vaccination and the duration of follow-up

Exclusion Criteria: The participant may not enter the trial if ANY of the following apply:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant skin disorder (psoriasis, contact dermatitis etc.), cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the PI or other delegated individual.
* Weight-for-age Z score of less than -3 or other clinical signs of malnutrition.
* History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunisation.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Sickle cell disease.
* Clinically significant laboratory abnormality at grade 2 or above as judged by the PI or other delegated individual.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Receipt of any vaccine in the 14 days preceding enrolment, or planned receipt of any other vaccine within 28 days following each study vaccination.
* History of vaccination with another malaria vaccine.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Known maternal HIV infection (no testing will be done by the study team).
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (for corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day; inhaled and topical steroids are allowed).
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

The following adverse events associated with vaccine immunisation constitute absolute contraindications to further administration of vaccine. If any of these events occur during the study, the participant must be withdrawn and followed until resolution of the event, as with any adverse event:

• Anaphylactic reaction following administration of vaccine.

The following adverse events constitute contraindications to administration of vaccine at that point in time; if any one of these adverse events occurs at the time scheduled for vaccination, the participant may be vaccinated at a later date, or withdrawn at the discretion of the Investigator. The participant must be followed until resolution of the event as with any adverse event:

* Acute disease at the time of vaccination (acute disease is defined as the presence of a moderate or severe illness with or without fever or symptoms suggestive of possible COVID-19 disease). All vaccines can be administered to persons with a minor illness such as diarrhoea or mild upper respiratory infection without fever, i.e. axillary temperature < 37.5°C.
* Temperature of >37.5°C (99.5°F) at the time of vaccination.

Ages: 5 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: The primary efficacy outcome is clinical malaria, defined as the presence of axillary temperature ≥37.5°C and P. falciparum parasite density >5000 asexual forms/µL. | Clinical malaria will be assessed 6 months post final vaccination
  To assess the protective efficacy against clinical malaria of R78C with Matrix-M™, and the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™, in children living in a malaria-endemic area, for 6 months after the final vaccination.
  Primary case definition for clinical malaria:
  • Presence of axillary temperature ≥37.5°C and/or history of fever within the last 24 hours AND P. falciparum asexual parasitaemia > 5000 parasites/µL
  Secondary case definitions for clinical malaria:
  * Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND EITHER P. falciparum asexual parasitaemia >0 parasites/µL OR positive RDT
  * Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND P. falciparum asexual parasitaemia >20,000 parasites/µL
Safety: To assess the safety and reactogenicity of R78C, RH5.1 and R21 with Matrix-M™ by assessing solicited adverse events (AEs) in children living in a malaria-endemic area until 6 months after administration of the final dose of vaccine. | Day 0,1-6,28,29-34,98,99-104,126,127-132,154,155-160,182,183-188.
  The occurrence of solicited local and systemic reactogenicity signs and symptoms will be assessed for 7 days following each vaccination (day of vaccination and 6 subsequent days)
  Foreseeable adverse reactions following vaccination with RH5.1, R78C or R21 and Matrix-MTM adjuvant are:
  * Local reactions: pain, erythema, warmth, swelling
  * Systemic reactions: drowsiness, fever, irritability/fussiness, loss of appetite
  These AEs will be listed as 'solicited AEs' providing they occur within 7 days of the day of vaccination.
Safety: To assess the safety and reactogenicity of R78C, RH5.1 and R21 with Matrix-M™ by assessing unsolicited adverse events (AEs) in children living in a malaria-endemic area until 6 months after administration of the final dose of vaccine. | Day 0,1-6,14,28,29-34,42,56,98,99-104,112,126,127-132,140,154,155-160,168,182,183-188,196.
  The occurrence of unsolicited AEs will be assessed for 7 days following each vaccination (day of vaccination and 6 subsequent days).
  Unsolicited AEs' are AEs other than the foreseeable adverse reactions occurring within the first 7 days, or any AEs occurring after the first 7 days after vaccination.
  For every unsolicited AE, an assessment of the relationship of the event to the administration of the vaccine will be undertaken by the PI or the PI-delegated clinician. An intervention-related AE refers to an AE for which there is a possible, probable or definite relationship to administration of a vaccine. An interpretation of the causal relationship of the intervention to the AE in question will be made, based on the type of event; the relationship of the event to the time of vaccine administration; and the known biology of the vaccine therapy
Safety: To assess the safety and reactogenicity of R78C, RH5.1 and R21 with Matrix-M™ by assessing serious adverse events (SAEs) in children living in a malaria-endemic area until 6 months after administration of the final dose of vaccine. | Throughout study completion, an average of 1 year
  The occurrence of SAEs during the whole study duration.
  An SAE is an AE that results in any of the following outcomes, whether or not considered related to the study intervention:
  * Death.
  * Life-threatening event. This does not include an AE that, if it occurred in a more severe form, might have caused death.
  * Persistent or significant disability or incapacity.
  * Hospitalisation or prolongation of hospitalisation, regardless of length of stay, even if it is a precautionary measure for continued observation. Hospitalisation for a pre-existing condition that has not worsened unexpectedly does not constitute an SAE.
  * An important medical event that may, based upon appropriate medical judgment, jeopardise the volunteer and/or require medical or surgical intervention to prevent one of the outcomes listed above.
  * Congenital anomaly or birth defect.

SECONDARY OUTCOMES:
Immunogenicity:To assess the humoral immunogenicity of R78C with Matrix-M™, and the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™ in children living in a malaria-endemic area. | Blood samples for immunogenicity will be taken at Day -30 to 0, 0, 42, 56, 182, 196, 238, and 350.
  Humoral immunogenicity will be assessed from blood samples taken at various timepoints. Immunogenicity will be determined following the quantification of antigen-specific IgG antibody levels (µg/mL readout) over time, as well as by in vitro growth inhibition assays (GIA) against P. falciparum parasites using purified total IgG and a single-cycle pLDH readout assay.
Efficacy: To assess the protective efficacy against clinical malaria of R78C with Matrix-M™, in children living in a malaria-endemic area, for 3 months after the final vaccination | 3 months after the final vaccination
  The definition for clinical malaria is as follows:
  1. Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND EITHER P. falciparum asexual parasitaemia >0 parasites/µL OR positive RDT
     or
  2. Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND P. falciparum asexual parasitaemia >20,000 parasites/µL
  Efficacy will be determined following the comparison of mean parasite density in each study arm
Efficacy: To assess the protective efficacy against clinical malaria of the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™, in children living in a malaria-endemic area, for 3 months after the final vaccination | 3 months after the final vaccination
  The definition for clinical malaria is as follows:
  1. Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND EITHER P. falciparum asexual parasitaemia >0 parasites/µL OR positive RDT
     or
  2. Presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND P. falciparum asexual parasitaemia >20,000 parasites/µL
  Efficacy will be determined following the comparison of mean parasite density in each study arm
Efficacy: To assess the protective efficacy against asymptomatic P. falciparum infection of R78C with Matrix-M™, and the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™, in children living in a malaria-endemic area. | 2 and 6 months after administration of the final dose of vaccine
  This will be measured by looking at the following:
  * Proportion of participants in each study arm that show presence of parasite density >5000 asexual forms/µL as measured by quantitative reverse-transcriptase PCR (qRT-PCR) from 14 days to 2 and 6 months after administration of the final study vaccination PLUS presence of axillary temperature <37.5°C and absence of history of fever within the last 24 hours
  * Proportion of participants in each study arm that show presence of parasite density >0 asexual forms/µL as measured by qRT-PCR from 14 days to 2 and 6 months after administration of the final study vaccination PLUS presence of axillary temperature <37.5°C and absence of history of fever within the last 24 hours
  * Parasite density in those with >0 asexual forms/µL as measured by qRT-PCR from 14 days to 2 and 6 after administration of the final study vaccination PLUS presence of axillary temperature <37.5°C and absence of history of fever within the last 24 hours
Efficacy: To assess the protective efficacy against gametocytaemia of R78C with Matrix-M™, and the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™, in children living in a malaria-endemic area | 2 and 6 months after administration of the final dose of vaccine
  Protective efficacy against gametocytaemia will be assessed by measuring the proportion of participants in each study arm that show the presence of gametocytes >0 gametocytes/μL as measured by qRT-PCR from 14 days to 2 and 6 months after administration of the final study vaccination
Efficacy: To assess the protective efficacy of R78C with Matrix-M™, and the combination of RH5.1 with Matrix-M™ and R21 with Matrix-M™, against prevalent moderate or severe anaemia at 6 months after administration of the final dose of vaccine | 6 months after administration of the final dose of vaccine
  Prevalent severe anaemia is defined as a documented haemoglobin (Hb) level <5.0 g/dL.
  Prevalent moderate anaemia is defined as a documented Hb level <8.0 g/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, Principal Investigator — Institut de Recherche en Sciences de la Sante, Burkina Faso
Locations (1):
- Institut de Recherche en Sciences de la Sante - Clinical Research Unit of Nanoro (IRSS-URCN), Nanoro, Burkina Faso